CLINICAL TRIAL: NCT04957901
Title: The Value of Monitoring Circulating Cell DNA (ctDNA) in Pediatric Lymphoma: A Prospective, Multicenter Clinical Study
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhuo Zhang, Director of department of pediatric cancer,Principal Investigator,Clinical Professor, Sun Yat-sen University
Other Study IDs: cDNA
Record Dates: First submitted 2021-07-05; First posted 2021-07-12 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-04

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Pediatric lymphoma protocol — The tumor tissue (FFPE) and plasma samples (bone marrow or cerebrospinal fluid samples if necessary) from the newly diagnosed patients were collected and sequenced by 475 genes panel before, during and post treatment.

SUMMARY:
The next-generation sequencing (NGS) based on liquid biopsy has been an emerging technology to identify tumor-specific genetic aberrations in malignant tumors. The tumor tissue (FFPE) and plasma samples from the newly diagnosed pediatric lymphoma patients were collected and sequenced by 475 genes panel before, during and post treatment, to evaluate the significance of the ctDNA in efficacy prediction, predicting recurrence or mechanism of resistance to chemotherapy for pediatric lymphoma.

DETAILED DESCRIPTION:
This is a prospective, multi-center, observational cohort study. The tumor tissue (FFPE) and plasma samples (bone marrow or cerebrospinal fluid samples if necessary) from the newly diagnosed patients were collected and sequenced by 475 genes panel before, during and post treatment. Collection and analysis the results of ctDNA and chemotherapy response, to explore the mutation map of pediatric lymphoma and to evaluate the significance of liquid biopsy for efficacy prediction, predicting recurrence, mechanism of resistance to chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Children with pediatric lymphoma (HL and NHL) that met the criteria and required treatment upon histological and pathological diagnosis;
2. Age: < 18 years old;
3. The working status of the Eastern Cooperative Oncology Group (ECOG) (PS) : 0-2 points;
4. CT/MRI measurable lesion was defined as the longest diameter of at least 1 lymph node ≥ 1.5cm, and it was clearly measurable in 2 vertical directions;
5. Complete clinical laboratory examination and pathological examination information;
6. Patients can be evaluated on time, and the required samples can be obtained throughout the testing process;
7. After the patient is informed of the project, the informed consent signed by the patient or his legal representative is obtained.

Exclusion Criteria:

* Patients with any of the following items will not be enrolled in this study:

  1. Incomplete baseline samples (preoperative plasma samples, tissue, bone marrow, cerebrospinal fluid) due to various reasons;
  2. The follow-up samples cannot be obtained during the monitoring process;
  3. The researcher considered it unsuitable for enrollment.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Asian population predominates
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The mutation rate of the ctDNA of pediatric lymphoma | From the beginning of observation to the end of observation（6 weeks) of the last enrolled patient

CONTACTS AND LOCATIONS:
Overall Officials: Yizhuo Zhang, Principal Investigator — Sun Yat-sen University CancerCenter
Locations (1):
- Yizhuo Zhang, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No